CLINICAL TRIAL: NCT00696150
Title: Can the Use of Ultrasound to Guide the Insertion of a Needle for an Anterior Psoas Compartment Nerve Block Increase Its Efficacy in Comparison to Traditional Techniques Utilising Loss of Resistance and Nerve Stimulation?
Brief Title: Can the Femoral Nerve Block be Improved by Ultrasound Guidance?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Golden Jubilee National Hospital (Other Government)
Responsible Party: Dr Erica Packard, NHS Greater Glasgow and Clyde health board
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ultrasound for hip # study-1; CSO reference CAF/07/05
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Pain
Keywords: ultrasound; hip; pain
MeSH Terms: conditions — Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- loss of resistance (Placebo Comparator): Anterior psoas compartment nerve block inserted using loss of resistance
  Interventions: Procedure: loss of resistance
- nerve stimulator (Active Comparator): Anterior psoas compartment nerve block inserted using nerve stimulator
  Interventions: Procedure: determination of method with highest efficacy (ultrasound or nerve stimulator); Procedure: nerve stimulator
- ultrasound (Active Comparator): Anterior psoas compartment nerve block inserted using ultrasound
  Interventions: Procedure: determination of method with highest efficacy (ultrasound or nerve stimulator)

INTERVENTIONS:
Procedure: determination of method with highest efficacy (ultrasound or nerve stimulator) — Use of ultrasound to guide the insertion of anterior psoas compartment block
  Arms: nerve stimulator; ultrasound
Procedure: nerve stimulator — The use of the nerve stimulator to guide insertion of the anterior psoas compartment block
  Arms: nerve stimulator
Procedure: loss of resistance — Use of ultrasound to guide the insertion of anterior psoas compartment block
  Arms: loss of resistance

SUMMARY:
Studies have suggested a link with effective pain relief and reduced illness and death in very unwell patients. This study will determine the most effective method of injecting local anaesthetic around the nerves which supply the hip joint. Local anaesthetic will be injected around the hips nerve supply using either ultrasound, loss of resistance or electrical nerve stimulator to guide the positioning of the needle on patients due for elective total hip replacement. The patient will then be observed for 30 minutes and the patient ability to move or feel the upper leg will recorded. A standard anaesthetic and a hip replacement operation will then be performed. Standard pain relief protocols will be used the operation and after the operation. After the operation we will record the amount of morphine used and how happy the patients have been with their treatment at 6 hours after the operation and at 24 hours after the operation. The first day the patient is able to walk on their new hip replacement will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary total hip arthroplasty under general anaesthesia
* ASA<=4
* Able to give informed consent
* Able to cooperate with sensory and motor testing of lower limb function

Exclusion Criteria:

* Abnormal clotting screen (coagulopathy) or thrombocytopenia (<100,000)
* Acute mental test score of <=7 at any time pre or post operatively
* Allergy to local anaesthetic
* Signs, symptoms or laboratory evidence of local infection or systemic sepsis
* No pre-existing neurological deficit (sensory or motor) affecting lower limb
* Patients with lower limb amputations

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with effective regional analgesia | Induction of anaesthesia

SECONDARY OUTCOMES:
hospital mortality | 1months after operation
sensory function in lateral cutaneous nerve | 0mins, 10mins 20mins post insertion of local anaesthetic
sensory function of femoral nerve | 0mins, 10mins, 20mins after insertion of local anesthetic
sensory function of obturator nerve | 0mins, 10mins, 20mins after insertion of local anesthetic
motor function of obturator nerve | 0mins, 10mins and 20minutes after insrtion of local anesthetic
motor function of femoral nerve | 0mins,10mins and 20mins post insertion of local anesthetic
acute mental test scores | 6hours and 24 hours post operatively
total morphine dose administered | 6hours and 24 hours post operstively
day first mobilise post operatively | post operatively 0-10 days
patient satisfaction scores | 6 hours and 24hours post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm watson, MB ChB FRCA, Study Chair — NHS Greater Glasgow and Clyde
Locations (4):
- United Kingdom (4):
  - Gartnavel General hospital, Glasgow, Lanarkshire
  - Glasgow Royal Infrimary, Glasgow, Lanarkshire
  - Golden Jubilee hospital, Glasgow, Lanarkshire
  - Royal alexandra hospital, Paisley, Renfrewshire